CLINICAL TRIAL: NCT04644367
Title: The Effects of a Biomechanical Based Tai Chi Intervention Program on Postural Stability and Gait in People With Parkinson's Disease
Brief Title: Effects of a Biomechanical-based Tai Chi Program on Gait and Posture in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Nok-Yeung Law, Principle Investigator, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-01-19-2284
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Gait; postural stability; falls; Tai Chi
MeSH Terms: conditions — Parkinson Disease | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: A prospective, single-blind, randomized control trial of 40 individuals with early-stage PD (Hoehn & Yahr stages 1 to 3).
Who Masked: Outcomes Assessor
Masking Description: The principle investigator, co-investigators will analyze and interpret the data, but will be blinded to the group allocation (single-blind). The principle investigator, co-investigators will restrict discussion of the study's outcomes with the research assistants who will be aware allocation, and who will be involved in data entry or collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi group (Experimental): The Tai Chi (TC) group will receive or be taught TC in a class size consisting of about 5-12 students. Classes will be taught by a TC master with more than 4 years of experience practicing either Yang or Wu style TC. The participants will be allowed to practice TC at home and during their leisure time so long as they keep an activity log of their daily TC practice. This monitoring form (i.e. activity log or journal) will be distributed to all members of this group and collected weekly.
  Interventions: Other: Tai Chi intervention
- Regular Physical Activity (control) group (Active Comparator): The regular physical activity (control) group will be asked to maintain or engage in at least 60 minutes of regular physical activity on their own for three times per week. The participants will be instructed as to the type of regular PA that they may engage in. These types of PA include: walking, cleaning or performing chores inside the home, and/or climbing the stairs. No restriction will be made to limit others forms of physical activity; individuals in the control group will be permitted to engage in organized sports, instructor-led class such as boxing, dance, etc. to ensure the participant recruitment process is feasible. Similar to the TC group, participants in this group will be asked to complete an activity log (or journal) that will be collected weekly to monitor their regular PA levels.
  Interventions: Other: Regular Physical Activity (control) group

INTERVENTIONS:
Other: Tai Chi intervention — TC classes will be 60 minutes long, offered three times per week over a 12-week period. The participants who receive the TC intervention will be encouraged to attend at minimum two of the three sessions offered per week. The TC classes will follow the same order that will begin with a 5 to 10 minutes warm up, 40 minutes of core activities, and 5 minutes of cool-down. The training intensity and difficulty level of the TC program will gradually proceed from low, moderate, to advance. The classes will be offered in a group setting at a convenient location within a community centre or gymnasium. Alternatively, classes will be offered outdoors in the park or by the canal during the spring-summer months. Due to the COVID-19 situation, additional adaptive measures will be taken using online social platforms such as ZOOM or Hangout to deliver the classes.
  Arms: Tai Chi group
Other: Regular Physical Activity (control) group — Regular Physical Activity group who will not be receiving the TC intervention
  Arms: Regular Physical Activity (control) group

SUMMARY:
Parkinson's disease (PD) is associated with changes in gait and posture that can lead to a higher frequency of falls and injuries in this population. Research has shown a positive effect of tai chi (TC) training on the movement capacity for those with PD, however the understanding of the impact of TC training on gait and postural stability in PD is lacking. This study aims to examine the impact of a biomechanical-based TC intervention on dynamic postural stability and how it relates to walking performance. It is hypothesized that the effects of the TC intervention will help to improve measures relating to postural stability, gait, and cognition.

DETAILED DESCRIPTION:
A prospective, single-blind, randomized control trial of 40 individuals with early-stage PD (Hoehn & Yahr stages 1 to 3). Those with PD will be randomly assigned to either a TC group or a control group. The TC group will participate in a biomechanical-based TC training program that is formed based on the movement analysis of TC and will be practiced two to three times a week for 12 weeks. The control group will be asked to engage or maintain their regular physical activity for a period of 12 weeks. The primary and secondary outcomes will be assessed at baseline, 6-week, and 12-week after commencing the study protocol. The primary outcome measures will include gait speed, cadence, step length during level surface walking (simple task) and fixed-obstacle crossing (challenging task); the dynamic postural stability will be indicated by the center of mass and center of pressure (COM-COP) separation distance and clearance distance measured during fixed-obstacle crossing. The secondary measures will be the Unified Parkinson's disease Rating scale (UPDRS-III), single leg-stance test with eyes open and closed, and three cognitive scores (Stroop Test, Trail Making Test- Part B, and the Wisconsin Card Sorting Test).

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with PD and demonstrate a disease severity ranging from 1 to 3 on the Hoehn and Yahr (H&Y) scale
* Have no fluctuations in motor symptoms as reported by the motor section of the Unified Parkinson's Disease Rating Scale (UPDRS-III)
* Have stable PD (such as levodopa or carbidopa) and doctor-prescribed medication use, that is, fluctuation did not occur at the time of medication intake;
* Can stand and walk independently
* Availability: three times per week over a period of 12 weeks
* Be able to engage in PA for at least 60 min on their own, thrice per week, without prior experience practicing TC regularly.

Exclusion Criteria:

* Enrolled into any other behavioral or pharmacological studies
* Have a Montreal Cognitive Assessment (MoCA) score of < 26/27 (that indicate some mild cognitive impairment (MCI))
* Have had a serious medical condition or uncontrolled hypertension (equal or greater than a systolic 180 or diastolic 110 reading)
* Have any debilitating conditions that could prevent them from performing any PA for a minimum of 60 minutes.
* Have practiced or have experience of practicing TC in an organized class or program within the last 5 years at the start of participation in the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Center of Mass-Center of Pressure (COM-COP) Separation Distance | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  The COM-COP separation distance will be determined from the 3D-motion capture data. The participants will be asked to walk at a self-selected/comfortable pace and to crossover a 20-centimeter-high obstacle placed in the middle of the walkway (5 trials; averaged reported in meters).
Change in Clearance Distance Height | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  The clearance distance of the toe and heel will be determined from the 3D-motion capture data. The participants will be asked to walk at a self-selected/comfortable pace and to crossover a 20-centimeter-high obstacle placed in the middle of the walkway (5 trials; averaged reported in centimeters). This distance will be determined by the marker position of the heel/toe away from the top of the obstacle.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | baseline
  The participants will be administered a set of instructions and be asked to perform a series of cognitive and motor tasks. The total time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points.
Change in Balance, Lower-limb Muscle Strength | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Balance and lower-limb muscle strength will be assessed using the Single-leg Stance Test with Eyes Open (SLO) and Closed (SLC). The participant will be asked to stand for as long as possible up to 60 seconds, with either eyes open or closed. Trials will be terminated if the participant loses his or her balance, or if his or her feet are moved from the initial position (randomized order; 3 trials; averaged time of trials reported in second).
Change in Mobility | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Mobility will be assessed using the Timed Up and Go (TUG) test. The participants will be instructed to stand up from a chair, walk 3 meters as quick and safely as possible, cross a line marked on floor, turn around, walk back, and sit down (3 trials; time of each trial recorded in seconds).
Change in Mental Flexibility | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Mental flexibility will be assessed using the Wisconsin Card Sorting Test (WCST). The participants will be given a deck of 64-cards and will be asked to sort the cards by shape, color, or number. The number of errors made, and number of successful sorted categories (maximum of 6) will be recorded (3 trials; number of errors made recorded).
Change in Processing Speed | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Processing speed will be assessed using the Trail Making Test Part B (TMT-B). The participants will be given a set of numbers and letters that they will be asked to connect with lines the numbers to letters in ascending order. The time that it takes the participant to complete this task will be recorded (3 trials; completion time of each trial recorded in seconds).
Change in Mental Switching | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Mental switching will be assessed with the Stroop Test. The participants will be asked to name the color but not to read the word on a card. A color-word score will be given based on the total correct identification of the correct color within 45 seconds (3 trials; the total score scored out of 40).
Change in Walking Speed | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Walking speed will be determined from the 3D-motion capture data collected along an 8-meter-long walkway. The participants will be asked to walk along the walkway at self-selected/comfortable pace (5 trials; averaged reported in m/s).
Change in Walking Cadence | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Walking cadence will be determined from the 3D-motion capture data collected along an 8-meter-long walkway. The participants will be asked to walk along the walkway at self-selected/comfortable pace (5 trials; averaged reported in steps or cycles/min).
Change in Walking Step Length | baseline, 6 weeks (mid-intervention), and 12 weeks (post-intervention)
  Step length will be determined from the 3D-motion capture data collected along an 8-meter-long walkway. The participants will be asked to walk along the walkway at self-selected/comfortable pace (5 trials; averaged reported in meters).

CONTACTS AND LOCATIONS:
Locations (1):
- Human Movement Biomechanics Laboratory, Ottawa, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Law NY, Li JX, Zhu Q, Nantel J. Effects of a biomechanical-based Tai Chi program on gait and posture in people with Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2023 Jun 30;24(1):241. doi: 10.1186/s13063-023-07146-x. PMID 37386473
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886